CLINICAL TRIAL: NCT03728062
Title: Mindfulness Meditation vs. Physical Exercise as Internal Recovery Strategies: Study on Comparative Effects on Stress, Fatigue, Burnout, Sleep Quality and Immunocompetence. A Randomized Controlled Trial
Brief Title: Mindfulness Meditation Versus Physical Exercise: Comparing Effects on Stress and Immunocompetence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Collaborators: Universidad Rey Juan Carlos (Other); Universidad de Zaragoza (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 0709201711717
Record Dates: First submitted 2018-10-11; First posted 2018-11-01 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-07

CONDITIONS: Stress; Health Knowledge, Attitudes, Practice
Keywords: Mindfulness; Physical exercise; Salivary Immunoglobulin A; Recovery strategy from stress
MeSH Terms: conditions — Behavior; Motor Activity | interventions — Mindfulness; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness meditation during lunch break (Experimental): Participants performed mindfulness meditation during lunch break at work place for a month, beginning with 15 minutes and ending with 30 minutes. They had available a "quiet room" and mp3 audios with guided meditations based on the MBSR program.
  Interventions: Behavioral: Mindfulness meditation
- Physical exercise during lunch break (Experimental): Participants performed physical exercises during lunch break at a gym for a month, beginning with 15 minutes and ending with 30 minutes. They were instructed to do cardio exercise such as running through a park or going to the gym for running, rowing, cycling or elliptical exercise. 20-140 beats per minute must be reach.
  Interventions: Behavioral: Physical exercise
- Control group (No Intervention): Participants continue their normal lunch routine.

INTERVENTIONS:
Behavioral: Mindfulness meditation — Guided mindfulness meditation focused on breath sensations, thoughts and emotions.
  Other Names: Mindfulness based intervention (MBSR)
  Arms: Mindfulness meditation during lunch break
Behavioral: Physical exercise — Cardio exercise at gym like rowing, eliptical, cycling, or running outside.
  Other Names: Cardio exercise
  Arms: Physical exercise during lunch break

SUMMARY:
The objective of this research project is to examine if including mindfulness meditation or physical exercise at lunch break improve workers' recovery from work stress. Therefore, 72 workers included either mindfulness meditation or physical exercise during their lunchbreaks for a month in order to find out if these recovery strategies have more favorable outcomes than usually spent lunch breaks concerning: a) psychological detachment, b) perceived stress, c) general health, d) burnout, e) fatigue, f) quality of sleep, g) cortisol awakening response and h) immunocompetence.

DETAILED DESCRIPTION:
The investigators conduct an intervention study in a sample of 72 knowledge-workers, who engaged in mindfulness meditation or physical activities for five weeks. They performed from 15 to 30 minutes during their lunch breaks. The investigators randomly assigned participants to three experimental conditions: 1) mindfulness meditation, 2) physical activity, 3) control group (lunch break as usual). Online questionnaires before and after intervention assessed long term changes regarding recovery processes, perceived stress, health, mindfulness and burnout. For daily changes, a mobile application was developed to assess changes once per day immediately after work. The investigators also collect saliva samples to map cortisol and immunoglobulin A excretion across the intervention period. The investigators had two follow-up measures one and six months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Knowledge-workers of an specific company with similar stress level.

Exclusion Criteria:

* Serious illness
* Regular meditation
* Regular physical exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Spanish version of the Perceived Stress Questionnaire of Levenstein | 8 months
  Validation of the Spanish version of the Perceived Stress Questionnaire of Levenstein et al. (1993). It is a scale to measure stress in psychosomatic disorders. It consists of 30 items, with Likert responses from 1(almost never) to 4 (almost always). The Spanish version has 6 factors: Harrassment-social acceptance, Overload, Irritability-tension-fatigue, Energy-Joy, Fear-anxiety, Self-realization-satisfaction. The higher score, the higher perceived stress.
Recovery Experience Questionnaire (Sonnentag et al., 2007) | 8 months
  Recovery Experience Questionnaire (Sonnentag et al. 2007) is a measure for assessing recuperation from work. It has 16 items divided into four subscales: psychological detachment, relaxation, mastery and control. Each subscale has 4 items. Every items has a 5-point scale from 1 (I do not agree al all) to 5 (I fully agree). Higher scores indicates a higher degree of recovery from work stress.
Spanish version of the General Health Questionnaire (Goldberg et al., 1997) | 8 months
  Short version of General Health questionnaire. It has 12 items divided into three subscales: Stress, Coping strategies and Self-steem. Every item has a Likert scale to answer from 0 to 3. Higher scores indicates worse general health.
Salivary Immunoglobulin A | 1 months
  Level changes from Baseline to 1 month follow-up. Samples were collected in Salivettes -trademark- (a plastic tube with a swab) twice a day: in the morning (round 7am) and after work (round 7pm). There were collected two Salivettes every of the three moment of measuring (pretest, postest and 1 month follow-up). That means there were taken 6 tubes for every participant.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Santed Germán, PhD, Study Director — Universidad Nacional Española a Distancia; Carlos María Alcover de las Heras, PhD, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Telefonica S.A, Telecom company, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sonnentag S, Venz L, Casper A. Advances in recovery research: What have we learned? What should be done next? J Occup Health Psychol. 2017 Jul;22(3):365-380. doi: 10.1037/ocp0000079. Epub 2017 Mar 30. PMID 28358572
- [Background] Bliese PD, Edwards JR, Sonnentag S. Stress and well-being at work: A century of empirical trends reflecting theoretical and societal influences. J Appl Psychol. 2017 Mar;102(3):389-402. doi: 10.1037/apl0000109. Epub 2017 Jan 26. PMID 28125263
- [Background] Sonnentag S, Arbeus H, Mahn C, Fritz C. Exhaustion and lack of psychological detachment from work during off-job time: moderator effects of time pressure and leisure experiences. J Occup Health Psychol. 2014 Apr;19(2):206-16. doi: 10.1037/a0035760. Epub 2014 Mar 17. PMID 24635737
- [Background] Nagel IJ, Sonnentag S. Exercise and sleep predict personal resources in employees' daily lives. Appl Psychol Health Well Being. 2013 Nov;5(3):348-68. doi: 10.1111/aphw.12014. Epub 2013 Oct 8. PMID 24395817
- [Background] Hahn VC, Binnewies C, Sonnentag S, Mojza EJ. Learning how to recover from job stress: effects of a recovery training program on recovery, recovery-related self-efficacy, and well-being. J Occup Health Psychol. 2011 Apr;16(2):202-16. doi: 10.1037/a0022169. PMID 21463049
- [Background] Sanz-Vergel AI, Sebastian J, Rodriguez-Munoz A, Garrosa E, Moreno-Jimenez B, Sonnentag S. [Adaptation of the "Recovery Experience Questionnaire" in a Spanish sample]. Psicothema. 2010 Nov;22(4):990-6. Spanish. PMID 21044543
- [Background] Hulsheger UR, Walkowiak A, Thommes MS. How can mindfulness be promoted? Workload and recovery experiences as antecedents of daily fluctuations in mindfulness. J Occup Organ Psychol. 2018 Jun;91(2):261-284. doi: 10.1111/joop.12206. Epub 2018 Mar 4. PMID 29861554
- [Background] Jamieson SD, Tuckey MR. Mindfulness interventions in the workplace: A critique of the current state of the literature. J Occup Health Psychol. 2017 Apr;22(2):180-193. doi: 10.1037/ocp0000048. Epub 2016 Sep 19. PMID 27643606
- [Background] Daubenmier J, Hayden D, Chang V, Epel E. It's not what you think, it's how you relate to it: dispositional mindfulness moderates the relationship between psychological distress and the cortisol awakening response. Psychoneuroendocrinology. 2014 Oct;48:11-8. doi: 10.1016/j.psyneuen.2014.05.012. Epub 2014 May 27. PMID 24971591
- [Background] Leicht CA, Goosey-Tolfrey VL, Bishop NC. Exercise intensity and its impact on relationships between salivary immunoglobulin A, saliva flow rate and plasma cortisol concentration. Eur J Appl Physiol. 2018 Jun;118(6):1179-1187. doi: 10.1007/s00421-018-3847-6. Epub 2018 Apr 7. PMID 29627864
- [Background] Kobayashi H, Song C, Ikei H, Park BJ, Kagawa T, Miyazaki Y. Diurnal Changes in Distribution Characteristics of Salivary Cortisol and Immunoglobulin A Concentrations. Int J Environ Res Public Health. 2017 Aug 31;14(9):987. doi: 10.3390/ijerph14090987. PMID 28858222
- [Background] Moreira A, Freitas CG, Nakamura FY, Drago G, Drago M, Aoki MS. Effect of match importance on salivary cortisol and immunoglobulin A responses in elite young volleyball players. J Strength Cond Res. 2013 Jan;27(1):202-7. doi: 10.1519/JSC.0b013e31825183d9. PMID 22395269